CLINICAL TRIAL: NCT05228054
Title: Treatment of Hemorrhoid With 1940nm Laser Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34
Record Dates: First submitted 2022-01-26; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids, laser, sclerotherapy
MeSH Terms: conditions — Hemorrhoids | interventions — Sclerotherapy

STUDY DESIGN:
Intervention Model Description: Patients with hemorrhoids 2-3st will be randomized in two groups
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser 1940nm (Experimental): Patients with hemorrhoidal deasease 2-3 st. who will be treated with laser 1940nm
  Interventions: Procedure: laser procedure
- sclerotherapy (Active Comparator): Patients with hemorrhoidal deasease 2-3 st. who will be treated with sclerotherapy
  Interventions: Procedure: sclerotherapy

INTERVENTIONS:
Procedure: laser procedure — In modified litothomy position patients with hemorrhoidal deasease will be treated with transcutaneous laser 1940nm 3watt in impulse regimen
  Arms: Laser 1940nm
Procedure: sclerotherapy — In modified litothomy position patients with hemorrhoidal deasease will be treated with sclerotherapy with Aethoxysklerol
  Arms: sclerotherapy

SUMMARY:
Patients with hemorrhoids 2-3 st will be treated with laser 1940nm or sclerothearapy with Aethoxysklerol

DETAILED DESCRIPTION:
Prospective randomized, control study. Patients with hemorrhoids 2-3 will be randomized in two groups. 100 patient in each. Patients will be treated with laser 1940nm or sclerothearapy with Aethoxysklerol.

Follow up for one year. Primary end point - recurrence of hemorrhoids desease.

ELIGIBILITY:
Inclusion Criteria:

hemorrhoids 2-3st

Exclusion Criteria:

Acute hemorrhoids IBD psychosomatic diseases previous surgical interventions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Reccurence rate | 12 months
  reccurence of hemorroids desease

SECONDARY OUTCOMES:
Pain intensity | 7 days
  Score representing patient's current pain intensity
  Minimum: 0 (no pain) Maximum: 100 (very severe pain)
QoL | 12 months
  The SF-36 is often used as a measure of a person or population's quality of life (QOL) The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia